CLINICAL TRIAL: NCT00978211
Title: Phase II Study of [90Y-DOTA]-TOC and [177Lu-DOTA]-TOC in Metastasized Neuroendocrine Tumors
Brief Title: DOTA-TOC in Metastasized Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAW002
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Neuroendocrine Tumors
Keywords: DOTATOC; somatostatin; radiopeptide; Yttrium; Lutetium; neuroendocrine; cancer
MeSH Terms: conditions — Neuroendocrine Tumors; Neoplasms | interventions — 1,4,7,10-tetraazacyclododecane- 1,4,7,10-tetraacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DOTA-TOC (Experimental): Treatment arm
  Interventions: Drug: DOTA-TOC Treatment

INTERVENTIONS:
Drug: DOTA-TOC Treatment — Intravenous injections of DOTA-TOC. Repeated treatment cycles for responders, except in case of
  * renal toxicity
  * loss of patient transferability or
  * denial of further treatment.
  Other Names: tetraazacyclododecanetetraacetic acid (DOTA) modified; somatostatin analog Tyr3-octreotide (TOC)

SUMMARY:
The investigators aim to explore the efficacy of [90Y-DOTA]-TOC and [177LuDOTA]-TOC therapy in advanced neuroendocrine cancer. Therefore, the investigators assess response, survival and long-term safety profile of systemic [90Y-DOTA]-TOC and [177LuDOTA]-TOC treatment in metastasized neuroendocrine cancer patients. Adverse events are assessed according to the criteria of the National Cancer Institute. Survival analyses are performed using multiple regression models.

DETAILED DESCRIPTION:
Background: Systemic treatment with the 90Yttrium (90Y) labeled, tetraazacyclododecanetetraacetic acid (DOTA) modified somatostatin analog Tyr3-octreotide (TOC) was introduced in 1998 (Otte et al. Lancet 1998). [90Y-DOTA]-TOC is administered intravenously and binds to the somatostatin receptor subtype 2, located on the surface of the tumor cell, and exerts its cytotoxic effects by β-irradiation. The treatment has moderate acute hematologic and nephrologic toxicity and has developed into a promising therapeutic tool for tumors expressing its target receptor (Iten et al. Clin Cancer Res 2007, Iten et al. Cancer 2009).

Study Aim: To explore the efficacy of [90Y-DOTA]-TOC and [177LuDOTA]-TOC therapy in advanced neuroendocrine cancer.

Study Hypothesis: Response to DOTA-TOC is correlated with prolonged survival.

Study Type: Clinical phase II, single-center, open-label trial

Patients: 1500 patients

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed neuroendocrine cancer
* stage IVc disease by definition of the American Joint Committee on Cancer, i.e. occurrence of distant metastases
* visible tumor uptake in the pretherapeutic somatostatin receptor subtype 2 scintigraphy (111In-Octreoscan)

Exclusion Criteria:

* concurrent anti-tumor treatment
* secondary malignancies
* pregnancy
* breast-feeding
* incontinence
* severe concomitant illness including severe psychiatric disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1499 (Actual)
Dates: Start 1997-09; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Response | 3 months

SECONDARY OUTCOMES:
Toxicity | 3 months
Survival | life-long

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Walter, MD, Dr., Principal Investigator — Institute of Nuclear Medicine; Inselspital Bern
Locations (1):
- University Hospital, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Otte A, Mueller-Brand J, Dellas S, Nitzsche EU, Herrmann R, Maecke HR. Yttrium-90-labelled somatostatin-analogue for cancer treatment. Lancet. 1998 Feb 7;351(9100):417-8. doi: 10.1016/s0140-6736(05)78355-0. No abstract available. PMID 9482300
- [Background] Iten F, Muller B, Schindler C, Rochlitz C, Oertli D, Macke HR, Muller-Brand J, Walter MA. Response to [90Yttrium-DOTA]-TOC treatment is associated with long-term survival benefit in metastasized medullary thyroid cancer: a phase II clinical trial. Clin Cancer Res. 2007 Nov 15;13(22 Pt 1):6696-702. doi: 10.1158/1078-0432.CCR-07-0935. PMID 18006770
- [Background] Iten F, Muller B, Schindler C, Rasch H, Rochlitz C, Oertli D, Maecke HR, Muller-Brand J, Walter MA. [(90)Yttrium-DOTA]-TOC response is associated with survival benefit in iodine-refractory thyroid cancer: long-term results of a phase 2 clinical trial. Cancer. 2009 May 15;115(10):2052-62. doi: 10.1002/cncr.24272. PMID 19280592
- [Derived] Marincek N, Jorg AC, Brunner P, Schindler C, Koller MT, Rochlitz C, Muller-Brand J, Maecke HR, Briel M, Walter MA. Somatostatin-based radiotherapy with [90Y-DOTA]-TOC in neuroendocrine tumors: long-term outcome of a phase I dose escalation study. J Transl Med. 2013 Jan 15;11:17. doi: 10.1186/1479-5876-11-17. PMID 23320604